# T.E.S.S® VERSION 2

Retrospective and Prospective, Multi centre Study on T.E.S.S® V2 Shoulder System

PROTOCOL No. ORTHO.CR.E13

**NCT NUMBER: NCT03431857** 

PROTOCOL VERSION: 2012-05-30 - Rev. 2.0

# **STUDY SPONSOR**

ZIMMER GMBH
SULZERALLEE 8
P.O. BOX
CH-8404 WINTERTHUR
SWITZERLAND

Title: Retrospective and Prospective, Multi centre Study on T.E.S.S® V2

Shoulder System

**Sponsor:** Zimmer GmbH

**Objectives:** The objective of this study is to evaluate mid-term (5-year) clinical

performance of the T.E.S.S® Version 2 Anatomic and Reverse prostheses in shoulder arthroplasty. Patient and Shoulder function will be collected along with Constant Score, radiographic and survivorship data.

Outcome

Measures

• Primary outcome:

- o Clinical efficacy using Constant Score
- Other outcome measures
  - Passive and active mobility
  - o Radiographic Evaluation
  - Complications (including dislocation and revisions/removals)
  - o Survivorship.

Indication/ Target Population: 200 subjects suitable for T.E.S.S® Shoulder Replacement can be included into this study: 100 subjects in each subgroup

# Inclusion/Exclusion criteria

#### Inclusion criteria

The inclusion criteria are the same as the indications stated in the G-Med cleared labeling for

the device.

The range of T.E.S.S.® shoulder prostheses are indicated in the following cases:

- Except in special cases, the "anatomic" type is indicated for:
  - Centered osteoarthritis of the shoulder
  - Humeral head fractures
  - Rheumatoid arthritis (with intact rotator cuff)
  - Avascular necrosis of the humeral head
- Except in special cases, the "reversed" type is indicated for:
  - Offset osteoarthritis of the shoulder
  - o Massive and non-repairable rotator cuff tears
  - Rheumatoid arthritis (with degenerative rotator cuff)
- Revision in cases of:
  - Replacement of an "anatomic" prosthesis with a "reversed" prosthesis
  - o Conversion of a hemi-arthroplasty into a total arthroplasty
  - o Increasing the size of the stem (length and/or diameter)
  - o Replacing a glenoid prosthesis
  - Replacing a competitor's prosthesis
  - In rare cases, removing a "reversed" prosthesis and replacing it with an "anatomic" prosthesis

# Additional inclusion criteria include

 Patient who read, understood study information and gave informed consent (oral or written depending on specific local regulatory requirements)

#### **Exclusion criteria**

The Exclusion criteria are the same as the indications stated in the G-Med cleared labeling for the device

### Contraindications:

Subjects displaying any of the following contra-indications shall be excluded from this evaluation:

- Local or systemic infections.
- Severe muscular, neurological, or vascular deficiency of the affected joint.
- Bone destruction or poor bone quality liable to affect the stability of the implant (Paget's disease, osteoporosis, etc.)
- Cases where the corolla cannot be two-thirds covered with bone stock and including the stem/corolla junction.
- Any concomitant complaint likely to affect the functioning of the implant.
- Allergy to any of the implant components.
- Local bone tumors.

Additional exclusion criteria include

• Patient over 18 under law supervision

## Length of Study:

The study assessment period will be 6,5 years: 18 months of recruitment and 5 years followup. The follow-up clinical reviews for all patients will be at discharge, 6 weeks, 6 months, 1 year, 2 years, 3 years, 4 years and 5 years.